CLINICAL TRIAL: NCT00897442
Title: Acquisition of Human Gynecologic Specimens to be Used in Studying the Causes, Diagnosis, Prevention and Treatment of Cancer
Brief Title: Collecting Tumor Samples From Patients With Gynecological Tumors
Status: Completed | Type: Observational
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Other Study IDs: GOG-0136; NCI-2009-00577 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); GOG-136; CDR0000078647; GOG-0136 (Other: NRG Oncology); GOG-0136 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Borderline Ovarian Clear Cell Tumor; Borderline Ovarian Serous Tumor; Cervical Adenocarcinoma; Cervical Adenosquamous Carcinoma; Cervical Small Cell Carcinoma; Cervical Squamous Cell Carcinoma, Not Otherwise Specified; Childhood Embryonal Rhabdomyosarcoma; Childhood Malignant Ovarian Germ Cell Tumor; Endometrioid Stromal Sarcoma; Gestational Trophoblastic Tumor; Malignant Mesothelioma; Malignant Ovarian Epithelial Tumor; Melanoma; Neoplasm of Uncertain Malignant Potential; Ovarian Brenner Tumor; Ovarian Clear Cell Cystadenocarcinoma; Ovarian Serous Cystadenocarcinoma; Paget Disease of the Vulva; Recurrent Cervical Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Ovarian Germ Cell Tumor; Recurrent Primary Peritoneal Carcinoma; Recurrent Uterine Corpus Carcinoma; Recurrent Vaginal Carcinoma; Recurrent Vulvar Carcinoma; Stage I Ovarian Cancer; Stage I Uterine Corpus Cancer; Stage I Vaginal Cancer; Stage I Vulvar Cancer; Stage IA Cervical Cancer; Stage IA Fallopian Tube Cancer; Stage IA Ovarian Cancer; Stage IA Ovarian Germ Cell Tumor; Stage IB Cervical Cancer; Stage IB Fallopian Tube Cancer; Stage IB Ovarian Cancer; Stage IB Ovarian Germ Cell Tumor; Stage IC Fallopian Tube Cancer; Stage IC Ovarian Cancer; Stage IC Ovarian Germ Cell Tumor; Stage II Ovarian Cancer; Stage II Uterine Corpus Cancer; Stage II Vaginal Cancer; Stage II Vulvar Cancer; Stage IIA Cervical Cancer; Stage IIA Fallopian Tube Cancer; Stage IIA Ovarian Cancer; Stage IIA Ovarian Germ Cell Tumor; Stage IIB Cervical Cancer; Stage IIB Fallopian Tube Cancer; Stage IIB Ovarian Cancer; Stage IIB Ovarian Germ Cell Tumor; Stage IIC Fallopian Tube Cancer; Stage IIC Ovarian Cancer; Stage IIC Ovarian Germ Cell Tumor; Stage III Borderline Ovarian Surface Epithelial-Stromal Tumor; Stage III Cervical Cancer; Stage III Uterine Corpus Cancer; Stage III Vaginal Cancer; Stage III Vulvar Cancer; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Ovarian Germ Cell Tumor; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Ovarian Germ Cell Tumor; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Ovarian Germ Cell Tumor; Stage IIIC Primary Peritoneal Cancer; Stage IV Borderline Ovarian Surface Epithelial-Stromal Tumor; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer; Stage IV Uterine Corpus Cancer; Stage IVA Cervical Cancer; Stage IVA Vaginal Cancer; Stage IVB Cervical Cancer; Stage IVB Vaginal Cancer; Stage IVB Vulvar Cancer; Uterine Corpus Cancer; Uterine Corpus Leiomyosarcoma; Vulvar Squamous Cell Carcinoma
MeSH Terms: conditions — Ovarian Germ Cell Cancer; Sarcoma, Endometrial Stromal; Gestational Trophoblastic Disease; Mesothelioma, Malignant; Melanoma; Brenner Tumor; Uterine Cervical Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tumor Samples

GROUPS / COHORTS (1):
- Ancillary-Correlative (biomarker sampling and analysis): Snap frozen tumor tissue, OCT molds of tumor tissue, formalin-preserved tumor tissue, buffy coat-prepared tumor tissue, and blood samples are collected and stored in the repository. Patient information is kept confidential, and patients are not informed of any research/test results from use of their tissues.
  Interventions: Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This laboratory study is collecting tumor tissue and blood samples from patients with gynecologic tumors. Collecting and storing samples of tumor tissue and blood from patients with cancer to study in the laboratory may help in the study of cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect gynecologic tissue and blood from participating Gynecologic Oncology Group (GOG) institutions.

II. To provide a repository for long-term storage of gynecologic tissue and blood that will be used in studies designed to better understand the molecular biology of gynecologic tumors.

III. To make available, through the GOG Tissue Bank, tissue and blood for proposed projects conducted by GOG and non-GOG investigators.

OUTLINE:

Snap frozen tumor tissue, OCT molds of tumor tissue, formalin-preserved tumor tissue, buffy coat-prepared tumor tissue, and blood samples are collected and stored in the repository. Patient information is kept confidential, and patients are not informed of any research/test results from use of their tissues.

ELIGIBILITY:
Inclusion Criteria:

* Any of the following:

  * Patients who have had gynecologic tissue removed during surgery to diagnosis, treat, monitor, and/or prevent primary, persistent, or recurrent gynecologic cancer of the ovary, peritoneum, fallopian tube, cervix, uterine corpus, vagina, or vulva, meeting at least one of the following criteria:

    * Group A: Women who underwent surgery, were diagnosed with a primary gynecologic malignancy of the ovary, cervix, uterine corpus, or vulva, and have primary tumor, normal tissue, and blood available for submission for this protocol

      * Patients with ovarian cancer including all stages, grades, and common epithelial cell types

        * Invasive cancers and serous and mucinous borderline tumors of low malignant potential are allowed
        * At least 1 gram of frozen primary tumor tissue must be submitted for this protocol for patients with FIGO stage III or IV epithelial ovarian cancer
      * Patients with an invasive malignancy of the cervix or uterine corpus including all stages, grades, and common cell types
      * Patients with squamous cell carcinoma of the vulva
    * Group B: Women who underwent surgery and were diagnosed with a rare gynecologic malignancy of the ovary, peritoneum, fallopian tube, cervix, uterine corpus, vagina, vulva, a gestational trophoblastic tumor, or a tumor arising in endometriosis, and have tumor tissue available for submission for this protocol

      * Patients with a rare gynecologic malignancy of the ovary including malignant germ cell tumors; sex cord-stromal tumors; malignant mixed mesodermal tumors; clear cell, mucinous, small cell, or transitional cell carcinomas; malignant Brenner tumors; or borderline tumors of low malignant potential (except serous and mucinous)
      * Patients with a rare gynecologic malignancy of the peritoneum, including primary peritoneal cancer or mesothelioma
      * Patients with carcinoma of the fallopian tube
      * Patients with a rare gynecologic malignancy of the cervix including verrucous, small cell, clear cell, serous, or adenoid cystic carcinomas; carcinoid tumors; malignant mixed mesodermal tumors; or leiomyosarcoma
      * Patients with a rare gynecologic malignancy of the uterine corpus including leiomyosarcoma; malignant mixed mesodermal tumors; endometrial stromal sarcomas; smooth muscle tumors of unknown malignant potential; or clear cell or small cell carcinomas
      * Patients with a rare gynecologic malignancy of the vagina including verrucous or clear cell carcinomas; melanoma; embryonal rhabdomyosarcoma; or endodermal sinus tumor
      * Patients with a rare gynecologic malignancy of the vulva including verrucous carcinoma; melanoma; aggressive angiomyxoma; sarcoma; malignant Paget's disease; or Bartholin gland carcinoma
      * Patients with a gestational trophoblastic tumor
      * Patients with a tumor arising in endometriosis
    * Group C: Women who underwent prophylactic oophorectomy and have at least 1 gram of ovarian tissue and blood available for submission for this protocol
    * Group D: Women who underwent surgery to monitor or treat a persistent or recurrent gynecologic malignancy of the ovary, peritoneum, fallopian tube, cervix, uterine corpus, vagina, or vulva, and have persistent or recurrent tumor, normal tissue, and blood available for submission for this protocol
* Concurrent primary cancers are allowed
* No benign cystic tumors of the ovary, including cystic epithelial tumors and mature cystic teratomas
* Prior cytotoxic chemotherapy allowed
* Prior hormonal therapy allowed
* Prior radiotherapy allowed
* Prior surgery allowed
* No more than 6 weeks after prior surgery

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients With Gynecological Tumors
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 1992-06; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Collection of gynecological tumor specimens and serum from patients at GOG institutions | Baseline
Create a repository for long-term storage of these specimens | Baseline
Make available tissue and blood for proposed projects | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cibull, Principal Investigator — NRG Oncology
Locations (187):
- United States (187):
  - Highlands Oncology Group PA - Fayetteville, Fayetteville, Arkansas
  - Washington Regional Medical Center - Fayetteville, Fayetteville, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Long Beach Memorial Medical Center-Todd Cancer Institute, Long Beach, California
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Olive View-University of California Los Angeles Medical Center, Sylmar, California
  - Colorado Gynecologic Oncology Group, Aurora, Colorado
  - University of Colorado Cancer Center - Anschutz Cancer Pavilion, Aurora, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Northside Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Our Lady Bellefonte Hospital, Ashland, Kentucky
  - Saint Elizabeth Medical Center South, Edgewood, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - Woman's Hospital, Baton Rouge, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - CHRISTUS Highland Medical Center, Shreveport, Louisiana
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - The Union Memorial Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Massachusetts Memorial Health Care, Worcester, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Gynecologic Oncology of West Michigan PLLC, Grand Rapids, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Saint Dominic-Jackson Memorial Hospital, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center, Kessler Air Force Base, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical CCOP, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - Pitt County Memorial Hosp Inc., Greenville, North Carolina
  - East Carolina University, Greenville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Akron General Medical Center, Akron, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates-Midtown, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Compass Oncology Rose Quarter, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Black Hills Obstetrics and Gynecology, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - East Tennessee State University, Johnson City, Tennessee
  - Southeast Gynecologic Oncology Associates, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - University Medical Center Brackenridge, Austin, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Clements University Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - The Methodist Hospital System, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Covenant Medical Center-Lakeside, Lubbock, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - MultiCare Auburn Medical Center, Auburn, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - MultiCare Good Samaritan Hospital, Puyallup, Washington
  - Virginia Mason CCOP, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Northwest NCI Community Oncology Research Program, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin